CLINICAL TRIAL: NCT06963944
Title: Investigation of the Relationship Between Physiological Dead Space and Intensive Care Unit Mortality in Mechanically Ventilated Adult Patients: A Prospective Observational Study
Brief Title: Physiological Dead Space and Intensive Care Mortality in Mechanically Ventilated Patients
Acronym: IRIS-MAP
Status: Completed | Type: Observational
Sponsor: Karadeniz Technical University (Other)
Responsible Party: Principal Investigator, A. Oguzhan KUCUK, MD, Assist. Prof., Karadeniz Technical University
Other Study IDs: 2024/154
Record Dates: First submitted 2025-04-20; First posted 2025-05-09 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-04

CONDITIONS: Invasive Mechanical Ventilation; Ventilation-Perfusion Mismatch; ICU Mortality; Critical Illness; End Tidal CO2
Keywords: Physiological Dead Space; Volumetric Capnography; Enghoff Equation; Mechanical Ventilation; ICU; Critical Care; Ventilation-Perfusion Mismatch; PaCO₂; EtCO₂; ICU Mortality; Gas Exchange; Respiratory Monitoring
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Mechanically Ventilated Adult ICU Patients: Adult patients (aged ≥18 years) who received invasive mechanical ventilation in a tertiary intensive care unit. All participants were prospectively monitored with volumetric capnography and arterial blood gas analysis to evaluate physiological dead space. No interventions were applied as part of the study.

SUMMARY:
This study investigates the relationship between physiological dead space and clinical outcomes, specifically mortality and discharge status, in adult patients receiving invasive mechanical ventilation in the intensive care unit (ICU). Physiological dead space refers to ventilated but non-perfused regions of the lungs and can be quantified using the Enghoff-modified Bohr equation based on capnographic and arterial CO₂ measurements.

While volumetric capnography is a valuable tool in anesthesiology and perioperative care, its use in ICU settings remains limited. By continuously monitoring physiological dead space at the bedside, this study aims to provide real-time insight into ventilation-perfusion mismatch and assess its prognostic significance in critically ill patients.

DETAILED DESCRIPTION:
Physiological dead space is defined as the portion of tidal volume that does not participate in effective gas exchange. It includes both anatomical and alveolar components and is a dynamic marker influenced by pulmonary perfusion, airway patency, ventilation settings, and lung pathology. In critically ill patients, particularly those receiving invasive mechanical ventilation, monitoring dead space may provide valuable insight into disease severity, ventilation-perfusion mismatch, and the adequacy of mechanical ventilation.

While capnography is routinely used in operating rooms and during anesthesia management, its role in intensive care units (ICUs) remains underutilized. Volumetric capnography offers a non-invasive, continuous method for assessing expired CO₂ and evaluating respiratory physiology in real time. Through the Enghoff-modified Bohr equation, physiological dead space can be calculated using the difference between arterial and end-tidal CO₂ (DS = (PaCO₂ - EtCO₂)/PaCO₂). This approach allows clinicians to quantify dead space without requiring invasive or complex instrumentation beyond standard ICU monitoring tools.

Previous research has identified an association between elevated dead space ventilation and increased mortality in conditions such as acute respiratory distress syndrome (ARDS), sepsis, and severe pneumonia. However, the utility of this parameter as a bedside prognostic tool in routine ICU practice remains limited by the lack of prospective validation and standardized monitoring protocols. Moreover, static measurements at a single time point may be insufficient to capture the clinical trajectory of critically ill patients, whereas trend analysis could provide more meaningful prognostic information.

This prospective observational study is designed to evaluate the relationship between physiological dead space and clinical outcomes, specifically ICU mortality and discharge disposition, in adult patients undergoing invasive mechanical ventilation. The study is conducted in a tertiary university hospital ICU and includes adult patients (≥18 years) who meet predefined inclusion criteria. Exclusion criteria are applied to eliminate potential confounders such as patients with noninvasive ventilation, pediatric cases, or those with significant technical limitations affecting capnographic measurements.

Data collection includes demographic characteristics, comorbidities, primary ICU admission diagnoses, ventilator parameters (tidal volume, PEEP, respiratory rate, minute ventilation, driving pressure), arterial blood gas values (PaO₂/FiO₂, PaCO₂), sedation level (RASS), vasoactive medication use, and daily volumetric capnography measurements (EtCO₂). Dead space values are recorded using standardized measurement windows, and time-series analysis is performed based on repeated observations during the ICU stay. The mode of discharge (survival, death, or transfer) is also documented.

The study aims to determine whether physiological dead space at ICU admission and its progression over time can serve as a reliable predictor of outcome. Additionally, it explores the feasibility of incorporating capnography-based dead space assessment into routine ICU monitoring as a noninvasive tool for early prognostication and ventilation optimization. Findings from this study may support broader use of volumetric capnography in intensive care medicine and contribute to individualized patient care strategies.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to the intensive care unit
* Receiving invasive mechanical ventilation
* Monitored with volumetric capnography and arterial blood gas analysis
* Informed consent obtained from legal representatives

Exclusion Criteria:

* Patients under 18 years of age
* ICU length of stay less than 24 hours
* Patient or legal representative refused participation
* Hemoglobin level < 7 g/dL
* Arterial PaCO₂ > 70 mmHg
* Signs of circulatory failure
* Lactate > 4 mmol/L
* Capillary refill time > 3 seconds
* PaCO₂ - Central venous CO₂ gradient > 8 mmHg (if applicable)
* Mean arterial pressure (MAP) < 65 mmHg
* Mottling score ≥ 2
* Body temperature > 38°C
* Arterial pH < 7.20
* Body mass index (BMI) > 40 kg/m²
* Carbon dioxide production (VCO₂) > 4 mL/kg

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consisted of adult patients (aged 18 years and older) who were admitted to a tertiary academic intensive care unit and required invasive mechanical ventilation for respiratory failure of various etiologies. All patients were managed in the ICU setting with advanced monitoring capabilities, including arterial blood gas analysis and volumetric capnography. Patients were enrolled consecutively during the study period based on predefined eligibility criteria. Individuals with hemodynamic instability, severe acidosis, or technical limitations preventing accurate dead space measurement were excluded. The study population reflects a critically ill cohort typically encountered in university hospital ICUs.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-04-19 (Actual); Study Completion 2025-04-19 (Actual)

PRIMARY OUTCOMES:
ICU Mortality | Up to ICU discharge day or 28 day
  All-cause mortality during the intensive care unit (ICU) stay.

SECONDARY OUTCOMES:
ICU Length of Stay | Through ICU stay, up to 28 days
  Number of days each patient spent in the ICU.
Mechanical Ventilation Duration | From initiation of invasive mechanical ventilation to extubation or death or, up to 28 days
  Total number of days under invasive mechanical ventilation.
Change in Physiological Dead Space Over Time | Daily measurements for up to 3 days in the ICU
  Temporal variation of physiological dead space calculated by Enghoff's modification of Bohr's equation (PaCO₂ - EtCO₂) / PaCO₂.
Relationship Between Physiological Dead Space and Oxygenation | Daily during ICU stay (up to 3 days)
  Correlation between dead space and oxygenation indices including PaO₂/FiO₂ ratio.

CONTACTS AND LOCATIONS:
Overall Officials: Mehtap Pehlivanlar Kucuk, MD, Assoc. Prof., Principal Investigator — Karadeniz Technical University, Faculty of Medicine
Locations (1):
- Karadeniz Technical University, Trabzon, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared due to privacy considerations and the lack of a formal data-sharing infrastructure for this study.